CLINICAL TRIAL: NCT01285440
Title: Determination of the Sensitivity of Low-dose Molecular Breast Imaging for the Detection of Small Breast Lesions
Brief Title: Use of Low-dose Molecular Breast Imaging for the Detection of Small Breast Lesions
Acronym: Lowdoseprebx
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie Hruska, Principal Investigator, Mayo Clinic
Other Study IDs: 10-000748
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Suspicious Breast Lesion for Which Biopsy is Scheduled
Keywords: breast; biopsy; suspicious lesion; molecular breast imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnostic Imaging

SUMMARY:
The purpose of this study is to show that improvements in the molecular breast imaging (MBI) technology will allow reduction of the administered dose of Tc-99m sestamibi while maintaining a sensitivity of 90% for tumor detection.

DETAILED DESCRIPTION:
A total of 150 patients will be studied. Each patient will have a suspicious lesion on mammogram, ultrasound or breast magnetic resonance imaging (MRI) for which biopsy is scheduled. The lesion size on mammogram, ultrasound or breast MRI must be less than 2 cm in diameter and must be considered "suspicious" or "highly suspicious" for malignancy. Following injection of 8 mCi Tc-99m sestamibi, all patients will undergo craniocaudal (CC) and mediolateral oblique (MLO) views of each breast using a molecular breast imaging (MBI) system incorporating the latest hardware and software algorithms. Each image will be acquired for 10 minutes in dynamic mode as 4 x 2.5 minute images. Summation of a given number of frames from each acquisition will yield images of an increasing mCi dose. Hence with an 8 mCi injection and a dynamic acquisition mode, we can evaluate the sensitivity of MBI as a function of administered doses of Tc-99m sestamibi ranging from 2 to 8 mCi. The thickness of the breast will be recorded to determine its relevance to lesion detectability.

Patient Selection

The goal of this study is to enroll 150 female patients in this study. The rationale for a study number of 150 patients is given in Appendix D. Patients referred for a mammogram, ultrasound or breast MRI study at Mayo Clinic Rochester will be considered for the study if they meet the following criteria:

* Have a lesion on mammogram, ultrasound or breast MRI that measured < 2 cm and is considered suspicious or highly suggestive of malignancy according to the Breast Imaging Reporting and Data System Atlas criteria (BI-RADS 4 or 5). (Note: while 2 cm is larger than the desired lesion size that we wish to study, this limit was recommended by our radiology colleagues as estimates of lesion size from mammography, ultrasound and MRI are not exact)
* Are scheduled for biopsy (needle and/or surgical biopsy) of the suspicious lesion
* Are > 18 years of age
* Had a negative pregnancy test or must be postmenopausal or surgically sterilized

Eligible patients will be offered enrollment if the time interval between mammogram, ultrasound or MRI and scheduled biopsy allows for performance of MBI. Patients with prior needle biopsy of the lesion will be excluded from this study, as such biopsies may effectively remove all or part of the lesion. Prospective patients will be identified by the radiologist based on findings in their mammographic, ultrasound or MRI studies.

ELIGIBILITY:
Inclusion Criteria:

-

Patients referred for a mammogram, ultrasound or breast MRI study at Mayo Clinic Rochester will be considered for the study if they meet the following criteria:

* Have a lesion on mammogram, ultrasound or breast MRI that measured < 2 cm and is considered suspicious or highly suggestive of malignancy according to the Breast Imaging Reporting and Data System Atlas criteria (BI-RADS 4 or 5). (Note: while 2 cm is larger than the desired lesion size that we wish to study, this limit was recommended by our radiology colleagues as estimates of lesion size from mammography, ultrasound and MRI are not exact)
* Are scheduled for biopsy (needle and/or surgical biopsy) of the suspicious lesion
* Are > 18 years of age
* Had a negative pregnancy test or must be postmenopausal or surgically sterilized

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 patients will be studied. Each patient will have a suspicious lesion on mammogram, ultrasound or breast MRI for which biopsy is scheduled. The lesion size on mammogram, ultrasound or breast MRI must be less than 2 cm in diameter and must be considered "suspicious" or "highly suspicious" for malignancy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Effective dose needed for detection of lesion | End of study when all data is collected
  The sensitivity of MBI for detection of the index lesion identified by other imaging will be determined as a function of the effective administered dose of Tc-99m sestamibi

CONTACTS AND LOCATIONS:
Overall Officials: Carrie B Hruska, PhD R-D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0